CLINICAL TRIAL: NCT06201585
Title: Single-port Robot-assisted Surgery for Gastric Cancer
Brief Title: Exploratory Study of Single-port Robot-assisted Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhao, Hebei Medical University, Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUTURE-05
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-port robot-assisted gastrectomy (Experimental): SHURUI Endoscopic Surgical Robotic System (SR-ENS-600)
  Interventions: Device: SHURUI Endoscopic Surgical Robotic System (SR-ENS-600)

INTERVENTIONS:
Device: SHURUI Endoscopic Surgical Robotic System (SR-ENS-600) — SHURUI Endoscopic Surgical Robotic System (SR-ENS-600)

SUMMARY:
This clinical study was a prospective, single-center, single-arm exploratory study. Subjects who meet the inclusion criteria will be enrolled in this study, where surgeons will perform single-port robot-assisted gastrectomy, and explore and evaluate the safety and efficacy of this clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and age ≤80 years old, regardless of gender;
2. patients who met the surgical indications and were confirmed by the investigator to be in need of laparoscopic surgery.
3. patients with American Society of Anesthesiologists (ASA) physical status classification ⅰ-ⅲ.
4. Be able to cooperate with the completion of visits and related examinations specified in the protocol.
5. Subjects voluntarily participated in the clinical trial and agreed or their guardians agreed to sign an informed consent.

Exclusion Criteria:

1. patients with severe heart, lung, brain, liver, or kidney diseases can not tolerate surgery or anesthesia;
2. those who cannot tolerate pneumoperitoneum;
3. patients with serious systemic diseases that are not suitable for surgical treatment according to the judgment of the investigator;
4. patients with a history of severe bleeding disease, hematopoietic dysfunction or coagulation dysfunction, who are not suitable for surgical treatment according to the judgment of the investigator, and long-term use of anticoagulant and antiplatelet drugs (antiplatelet aggregation drugs were discontinued less than 1 week before surgery);
5. patients with active pulmonary tuberculosis;
6. HIV antibody positive; Hepatitis B surface antigen (HbsAg) positive and hepatitis B virus DNA (HBV-DNA) copy number higher than the detection limit or normal range; Hepatitis C virus (HCV) antibody positive; Patients with positive treponema pallidum antibody and high risk of infection judged by the researcher;
7. with epilepsy, psychiatric history or cognitive impairment;
8. pregnant and lactating women;
9. Extensive and severe adhesion in the abdominal cavity caused the inability to perform puncture to establish pneumoperitoneum, and it was difficult to isolate and expose the lesion; A history of major abdominal surgery and abdominal radiotherapy were included, according to the investigator's judgment Situations where there is a risk of extensive adhesion;
10. participants who participated in other interventional clinical trials within 3 months before screening;
11. other circumstances that the investigator deemed inappropriate to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
The rate of intraoperative complications | The day of surgery
  Intraoperative complications, including organ injury and vascular injury, were evaluated
The rate of postoperative complications | Postoperative 30 days
  Postoperative complications, including postoperative bleeding, fever, and incisional infection, were evaluated using the Clavien-Dindo grading system to determine whether the occurrence of complications was related to the study instrument or surgery.

OTHER OUTCOMES:
Intraoperative system failure rate | The day of surgery
Surgical completion rate | The day of surgery
Intraoperative blood loss | The day of surgery
Operation time | The day of surgery
Preoperative device assembly time | The day of surgery
Intraoperative instrument operation error rate | The day of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Shijiazhuang, Hebei, China